CLINICAL TRIAL: NCT07346963
Title: Evaluation of Demographic, Clinical, and Healthcare Utilization Characteristics of Respiratory Syncytial Virus (RSV) Positive Cases Under 5 Years Presenting to Pediatric Emergency Departments in Türkiye: A Multicenter, Prospective Observational Study (TRUST-RSV)
Brief Title: RSV-Positive Children <5 Years Presenting to Pediatric Emergency Departments in Türkiye: TRUST-RSV
Acronym: TRUST-RSV
Status: Not yet recruiting | Type: Observational
Sponsor: Eskisehir Osmangazi University (Other)
Responsible Party: Principal Investigator, Emre Güngör, Emre Güngör, MD (Assistant Professor) , Principal Investigator, Eskisehir Osmangazi University
Other Study IDs: TRUST-RSV-v001; 2025-16 (Other: Eskisehir Osmangazi University Scientific Research Projects Unit)
Record Dates: First submitted 2025-12-17; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2025-12

CONDITIONS: Respiratory Syncytial Virus Infection; Acute Bronchiolitis Due to Respiratory Syncytial Virus; Pneumonia; Upper Respiratory Tract Infection
Keywords: pediatric emergency department; multicenter; prospective; healthcare utilization
MeSH Terms: conditions — Respiratory Syncytial Virus Infections; Pneumonia; Respiratory Tract Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Respiratory syncytial virus (RSV) is a leading cause of acute lower respiratory tract infection in infants and young children and contributes substantially to pediatric emergency department (ED) visits and hospitalizations. In Türkiye, nationally representative prospective data describing the epidemiology, clinical spectrum, and resource utilization of RSV-positive children presenting to pediatric EDs remain limited. This multicenter prospective observational study aims to characterize demographic and clinical features of RSV-positive children under 5 years of age presenting to participating pediatric EDs across two consecutive RSV seasons, and to quantify key healthcare utilization outcomes, including ED observation duration, hospitalization, and intensive care unit (ICU) admission.

DETAILED DESCRIPTION:
This is a multicenter, prospective observational cohort study conducted in pediatric emergency departments in Türkiye over a consecutive RSV season. Eligible participants are children younger than 5 years who present to a participating pediatric ED with at least one compatible clinical diagnosis and have RSV infection confirmed by a nasopharyngeal sample using either a rapid antigen test or PCR, based on local site capacity. Written informed consent will be obtained from a parent or legal guardian prior to study procedures.

Standardized case report forms will be used to collect demographics (age, sex, region, socioeconomic indicators), relevant risk factors (e.g., prematurity, congenital heart disease, chronic lung disease, passive smoke exposure, breastfeeding status), presenting symptoms, vital signs and physical examination findings, diagnostic evaluations (radiology and laboratory results as available), and clinical management and outcomes. Outcomes of interest include ED observation duration, disposition (discharge vs hospitalization), ICU admission, and, when applicable, the need for oxygen or ventilatory support. Data will be entered into a secure centralized database. The study will evaluate seasonal and regional patterns and will explore predictors of severe outcomes among RSV-positive children using multivariable models.

ELIGIBILITY:
Inclusion Criteria:

* Age <5 years at presentation
* Presentation during RSV season (2025-2026 )
* RSV infection confirmed from a nasopharyngeal sample by rapid antigen test or PCR according to site capacity
* Presentation to a participating pediatric ED with at least one of the following clinical diagnoses: upper respiratory tract infection, bronchiolitis, pneumonia, apnea, seizure/convulsion, or myocarditis
* Written informed consent obtained from a parent or legal guardian.

Exclusion Criteria:

* Parent or legal guardian declines consent

Ages: 28 Days to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The study population consists of children aged <5 years presenting to participating pediatric emergency departments in Türkiye during consecutive RSV season (2025-2026 ) who have respiratory syncytial virus (RSV) infection confirmed from a nasopharyngeal specimen using rapid antigen testing and/or PCR according to local site capacity and standard clinical practice. Eligible participants include RSV-positive children evaluated for compatible clinical diagnoses at presentation (e.g., upper respiratory tract infection, bronchiolitis, pneumonia, apnea, seizure/convulsion, or myocarditis). Enrollment requires written informed consent from a parent or legal guardian; children are excluded only if consent is declined. Clinical management is not assigned by the protocol and follows routine care; participants are observed for outcomes during the index emergency department encounter and, when applicable, through the index hospitalization.
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Hospitalization rate | Index ED visit (from ED presentation/triage to ED disposition decision and departure from the ED for inpatient admission or discharge), up to 24 hours.
  Proportion of children with laboratory-confirmed RSV infection presenting to participating pediatric EDs who are hospitalized from the index ED encounter. "Hospitalized" is defined as admission from the ED to an inpatient unit (ward) or intensive care unit (ICU) immediately following ED evaluation; children discharged home are classified as not hospitalized.
ICU admission rate among hospitalized RSV-positive children | During the index hospitalization, from hospital admission to hospital discharge, up to 24 hours.
  Proportion of hospitalized children with laboratory-confirmed RSV infection who require admission to an intensive care unit (ICU) at any time during the index hospitalization. ICU admission is defined as transfer from the ED or inpatient ward to an ICU for higher-level monitoring and/or organ support.
Need for respiratory support among RSV-positive children | From hospital admission to hospital discharge during the index hospitalization, up to 24 hours.
  Proportion of RSV-positive children who receive any respiratory support documented in the medical record, including supplemental oxygen (any delivery method) and/or noninvasive ventilation (e.g., HFNC/CPAP/BiPAP per local practice) and/or invasive mechanical ventilation.

SECONDARY OUTCOMES:
ED length of stay (ED observation duration) among RSV-positive children | Index ED visit (from ED arrival/registration or triage to ED disposition and ED departure), up to 24 hours.
  Time from ED arrival/registration (or triage time, per site practice) to ED disposition, defined as discharge home or departure from the ED for inpatient admission. Duration will be reported in hours.
Occurrence of RSV-associated complications during the index visit | From ED arrival to hospital discharge, up to 24 hours.
  Presence of pre-specified complications documented during the index ED visit and/or hospitalization (e.g., apnea requiring intervention, seizure/convulsion, myocarditis, suspected bacterial co-infection, or other clinically documented complications).
Diagnostic evaluations performed during the index visit | From ED arrival/registration (or triage) through hospital discharge for the index episode of care, up to 24 hours.
  Proportion of participants who undergo any diagnostic evaluation during the index visit as documented in the medical record and recorded in the study database. Diagnostic evaluations include, but are not limited to, chest radiography and laboratory testing performed in accordance with the standard of care.

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because the study was not designed with an IPD-sharing plan in place, and the current ethics approvals and informed consent documents do not include provisions for public IPD sharing.

REFERENCES:
- [Result] Tan L. A clinical observation on therapeutic effects of acupuncture for allergic rhinitis. J Tradit Chin Med. 1999 Jun;19(2):129-31. No abstract available. PMID 10681872
- [Result] Conti CR. Evolution of NCEP guidelines: ATP1-ATPIII risk estimation for coronary heart disease in 2002. National Cholesterol Education Program. Clin Cardiol. 2002 Mar;25(3):89-90. doi: 10.1002/clc.4960250302. No abstract available. PMID 11890375